CLINICAL TRIAL: NCT07219043
Title: A Double-Blind, Placebo-Controlled, Multicenter, Randomized Phase 2 Trial Evaluating the Efficacy and Safety of Felzartamab in Recipients of Kidney Transplants With Late Isolated Microvascular Inflammation (MVI)
Brief Title: A Study to Learn About the Effects of Felzartamab Infusions in Adults With Kidney Transplants Who Have Late Isolated Microvascular Inflammation
Acronym: TRANSPIRE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 299AR201; 2025-521742-15 (Other: EU CT Number)
Record Dates: First submitted 2025-10-17; First posted 2025-10-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Microvascular Inflammation
Keywords: Kidney Transplant; Kidney Transplant Rejection
MeSH Terms: interventions — felzartamab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a 2-part trial: Part A will be randomized and placebo-controlled, and Part B will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Felzartamab (Experimental): Participants will receive multiple IV doses of felzartamab.
  Interventions: Drug: Felzartamab
- Placebo and Felzartamab (Placebo Comparator): Participants will receive multiple IV doses of placebo followed by multiple doses of IV felzartamab.
  Interventions: Drug: Felzartamab; Drug: Placebo

INTERVENTIONS:
Drug: Felzartamab — Administered IV
  Other Names: MOR202, MOR03087, TJ202, HIB202, BIIB148
Drug: Placebo — Administered IV
  Arms: Placebo and Felzartamab

SUMMARY:
In this study, researchers will learn more about a drug called felzartamab in people who have received a kidney transplant and later developed a condition called microvascular inflammation (MVI). MVI is a type of injury to small blood vessels in the transplanted kidney and may be a sign of rejection by the body. It can lead to serious kidney problems over time.

The main goal of the study is to learn about the effect felzartamab has on inflammation in the transplanted kidney. The main question researchers want to answer is:

• How many participants have no signs of active inflammation in the transplanted kidney after 24 weeks of treatment with felzartamab?

Researchers will also study how felzartamab affects kidney function, immune activity, and overall health. They will monitor safety through kidney biopsies, lab tests, and by recording adverse events throughout the study.

Adverse events are unwanted health problems that may or may not be caused by the study drug.

The study will be done in 2 parts as follows:

* Participants will be randomly assigned to receive either felzartamab or a placebo. A placebo looks like the study drug but contains no real medicine.
* In Part A, participants will receive their assigned drug for 24 weeks. Neither the researchers nor the participants will know who is receiving felzartamab or placebo.
* Part B will last another 28 weeks. All participants will receive felzartamab and both participants and researchers will know this.
* All treatments will be given by intravenous (IV) infusion at the study site.
* Participants will have kidney biopsies at the start of the study, at week 24, and at week 52 to help measure changes in inflammation.
* Participants will stay in the study for about 1 year.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the efficacy of felzartamab compared to placebo in kidney transplant recipients diagnosed with complement activation (C4d)-positive or C4d-negative donor-specific antibody (DSA)-negative MVI (Part A). The secondary objectives of the study are to evaluate the efficacy of felzartamab compared to placebo through additional clinical endpoints (Part A), summarize safety and efficacy of felzartamab up to Week 52 in kidney transplant recipients diagnosed with C4d-positive or C4d-negative DSA negative MVI (Part B) and to assess the pharmacokinetic (PK) profile and immunogenicity of felzartamab (Parts A and B).

ELIGIBILITY:
Key Inclusion Criteria:

* C4d-positive or C4d-negative DSA-negative MVI (biopsy-confirmed) without T cell-mediated rejection (TCMR) per central reading, as defined by the Banff 2022 criteria.
* Biopsy must be within 3 months (preferably within 1 month) prior to randomization.

  a. For participants who received any prior treatment for antibody-mediated rejection (AMR), MVI, or TCMR as outlined in Exclusion Criterion 5, the biopsy must be performed at least 6 weeks after completing (or stopping) prior treatment.
* Kidney transplant at least 6 months prior to Screening visit (recipients of either living or deceased donors).
* DSA: Human leukocyte antigen (HLA) Class I and II antigen-specific DSA-negative (preformed and de novo DSA) as determined by the local laboratory's definition of positivity using single-antigen bead-based assays within 3 months prior to randomization.

Key Exclusion Criteria:

* Transplant: Blood type (ABO)-incompatible transplant.
* History of multiple organ transplants including en bloc and dual kidney transplants.
* Presence of HLA donor-specific antibodies.
* Acute, rapid decline in renal function, defined as a participant likely to require renal replacement therapy within the next 30 days as determined by the Investigator.
* Prior AMR or TCMR treatment (with the exception of corticosteroids) within 3 months prior to randomization is excluded as listed below. Participants who received any of these treatments between 3 and 6 months prior to randomization must have both a renal biopsy (IC3) and DSA testing at least 6 weeks after completing (or stopping) treatment in order to confirm continuing DSA-negative MVI and to determine eligibility:

  1. Intravenous or subcutaneous immunoglobulin (IVIg or subcutaneous immunoglobulin [SCIg]) or PLEX.
  2. Complement system inhibitors (e.g., eculizumab).
  3. Proteasome inhibitors (e.g., bortezomib).
  4. Tocilizumab.
  5. Any other investigational agent within 3 months or 5 half-lives (whichever is longer) of randomization.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2028-02-10 (Estimated); Study Completion 2028-02-10 (Estimated)

PRIMARY OUTCOMES:
Part A: Percentage of Participants Who Achieve Biopsy-proven Histologic Resolution (BPHR) | Week 24

SECONDARY OUTCOMES:
Part A: Microvascular Inflammation (MVI) Score | Week 24
Part A: Percentage of Participants Who Achieve an MVI Score of 0 | Week 24
Part A: Change from Baseline in Estimated Glomerular Filtration Rate (eGFR) | Baseline, Week 24
Part A: Percentage of Participants in the Complement Activation (C4d) Positive Cohort who Achieve BPHR | Week 24
Part B: Percentage of Participants Who Achieve BPHR | Weeks 24 and 52
Part B: MVI Score | Weeks 24 and 52
Part B: Percentage of Participants Who Achieve an MVI Score of 0 | Weeks 24 and 52
Part B: Change from Baseline in eGFR | Baseline, Weeks 24 and 52
Part B: Time to All-cause Allograft Loss | Up to Week 52
Parts A and B: Number of Participants with Adverse Events (AEs) | From first dose of study drug up to end of study follow-up (up to week 57)
Parts A and B: Percentage of Participants with T Cell-mediated Rejection (TCMR) by Biopsy | Weeks 24 and 52
Parts A and B: Number of Participants with Clinically Significant Laboratory Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Number of Participants with Clinically Significant Vital Signs Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Number of Participants with Clinically Significant Electrocardiogram (ECG) Abnormalities | From time of first dose to end of trial visit (Up to Week 52)
Parts A and B: Felzartamab Serum Concentration | Up to Week 52
Parts A and B: Number of Participants with Anti-drug Antibodies (ADAs) Against Felzartamab | Baseline, up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (3):
  - Cooperman Barnabas Medical Center, West Orange, New Jersey
  - The Ohio State University, Columbus, Ohio
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Hospital de Base da Faculdade de Medicina de São José do Rio Preto, Vila São José, São José Do Rio Preto, Brazil

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/